CLINICAL TRIAL: NCT01419639
Title: Phase II Study of Everolimus (RAD001) in Children and Adults With Neurofibromatosis Type 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Novartis Pharmaceuticals (Industry); The Children's Tumor Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD001 NF2 (11-00587); 2010-10-011 (Other Grant/Funding Number: Children's Tumor Foundation)
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Neurofibromatosis Type II
Keywords: Neurofibromatosis Type II; cranial nerve schwannomas; meningiomas; ependymomas
MeSH Terms: conditions — Neurofibromatosis 2; Meningioma; Ependymoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Experimental): RAD001 taken orally continuously until disease progression or unacceptable toxicity, dosed according to age
  Interventions: Drug: Everolimus (RAD001) , Afinitor®

INTERVENTIONS:
Drug: Everolimus (RAD001) , Afinitor® — Everolimus will be provided by Novartis. Everolimus is formulated as tablets for oral administration of 2.5 mg, 5 mg, 10 mg strength. Everolimus will be self-administered (by the patients themselves) or administered by the patient's parent or guardian (for minors). The investigator will instruct the patient to take the study drug exactly as specified in the protocol. Depending the age-based dosing schedule, everolimus should be administered orally once (or twice) daily, preferably in the morning (and evening), at the same time every day with our without food. Everolimus tablets should be swallowed whole with a glass of water. The tablets must not be chewed or crushed. In cases where tablets can not be swallowed, the tablets should be disintegrated in water just prior to being taken. Everolimus will be administered orally as per the age-based dosing schedule continuously from study day 1 until progression of disease or unacceptable toxicity.
  Other Names: Afinitor®

SUMMARY:
This trial studies whether Everolimus is efficacious in treating neurofibromatosis 2.

DETAILED DESCRIPTION:
Everolimus (RAD001) has been in clinical development since 1996 as an immunosuppressant in solid organ transplantation and has obtained marketing authorization (Certican®) for prophylaxis of rejection in renal and cardiac transplantation in a number of countries, including the majority of the European Union. Everolimus has been in development for patients with various malignancies since 2002. Everolimus 2.5mg, 5mg and 10mg tablets were approved under the trade name Afinitor® for patients with advanced renal cell carcinoma (RCC) after failure of treatment with Sutent® (sunitinib) or Nexavar® (sorafenib) in the US, EU and several other countries and is undergoing registration in other regions worldwide. Afinitor® was also recently approved for the treatment of patients with subependymal giant cell astrocytoma (SEGA) associated with tuberous sclerosis (TS) who require therapeutic intervention but are not candidates for curative surgical resection. Everolimus is being investigated as an anticancer agent based on its potential to act: 1. Directly on the tumor cells by inhibiting tumor cell growth and proliferation; and 2. Indirectly by inhibiting angiogenesis leading to reduced tumor vascularity.

For pediatric cancer patients, safety of RAD001 has been established in a phase 1 trial and the recommended phase II dose is 5 mg/m2 once daily. This existing pediatric data allows for inclusion of children in this phase 2 trial, which is an important consideration since some NF2 patients with the most aggressive clinical course present at school age.

RAD001 was recently approved by the Food and Drug Administration (FDA) for the treatment of children and adults with subependymal giant cell astrocytoma (SEGA), a benign brain tumor associated with tuberous sclerosis (TS). Although surgical resection is effective at tumor reduction, serious complications may follow a radical resection, such as permanent deafness and facial nerve damage. Most importantly, the tumors often recur after surgery. Radiation therapy (RT) has been proposed as an alternative. However, its safety and efficacy in the NF2 population has not been established. A medical therapy option is desperately needed. This study is a single-center, 2-stage, phase II open-label study. All subjects will get RAD001 taken continuously until disease progression or unacceptable toxicity. The primary objective of this study is to look at the objective response rate to RAD001 in patients with NF2-related tumors including cranial nerve schwannomas, meningiomas and ependymomas. Participation will consist of screening/baseline visit(s), Day 1, Weeks 1, 2, and 4; and up to 12 cycles and will include standard of care procedures such as medical history, vital signs, physical examinations, ECGs, MRIs, audiograms, and laboratory tests. Novartis will provide the RAD001 free of charge to eligible study subjects. The primary efficacy response for study purposes will be a greater than or equal to 15% reduction in tumor volume in any of the target tumors (partial response). Complete disappearance of any of the target tumors will constitute a complete response (CR).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 years and body surface area ≥ 0.5 m2
* Meets diagnostic criteria for NF2
* At least one volumetrically measurable and ≥ 0.5 cc NF2-related brain or spinal tumor (schwannoma, ependymoma, meningioma - histological confirmation not required) with radiographic evidence of progression (either as unequivocal progression on conventional MRI, or a >10% volume increase by 3D volumetrics) over the past ≤12 months, designated as the primary target tumor OR Volumetrically measurable and ≥ 0.5 cc VS with ipsilateral progressive hearing loss over the past ≤12 months, designated as the primary target tumor
* Progressive Hearing Loss Criteria for Enrollment: Audiogram showing drop in pure tone average (PTA) of 10dB HL at ≥ 2 nonconsecutive or consecutive frequencies or drop in speech discrimination score (SDS) below the 95% critical difference threshold, compared to previous audiogram ≤ 1 year prior.
* Karnofsky/Lansky performance status (PS) 50-100%. Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb > 9 g/dL
* Adequate liver function as shown by:

  1. serum bilirubin ≤ 1.5 x ULN
  2. ALT and AST ≤ 2.5x ULN
* INR ≤ 1.5. (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at time of enrollment.)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Fully recovered from acute toxic effects of any prior chemotherapy, biological modifiers or radiotherapy
* Any neurologic deficits must be stable for ≥ 1 week
* Able to provide signed informed consent (or consent by parent/legal guardian for minors)

Exclusion Criteria:

* Patients currently receiving medical anticancer therapies or who have received medical anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, antibody based therapy, etc.)
* Radiation therapy to a study target tumor within 1 year prior to enrollment, or any radiation therapy within 4 weeks prior to enrollment.
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  1. Symptomatic congestive heart failure of New York heart Association Class III or IV
  2. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  3. severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
  4. uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN (Note: Optimal glycemic control should be achieved before starting trial therapy.)
  5. active (acute or chronic) or uncontrolled severe infections
  6. liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).

Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.

* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes. (Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of everolimus)
* Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients who have received prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias A Karajannis, MD, MS, Principal Investigator — New York University
Locations (1):
- New York University Medical Center, New York, New York, United States

REFERENCES:
- See also: New York University Medical Center — http://www.med.nyu.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 people enrolled; a total of 9 completed study
Period: Overall Study
Arm/Group | RAD001
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | RAD001
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 27 [12 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response
Description: To estimate the objective response rates to RAD001 in patients with NF2-related tumors including cranial nerve schwannomas, meningiomas and ependymomas. Radiographic response for study purposes = greater than or equal to 15% reduction in tumor volume in any of the target tumors (partial response). Complete disappearance of any of the target tumors = complete response. MRI of the brain and spine will be performed every 3 months. If an objective response (15% reduction in tumor volume compared to baseline) is observed in any target tumor or stable disease, drug will be continued.
Time Frame: 1 Year
Measure: Number; unit: participants
Units Other Than Participants: Tumors
Arm/Group | RAD001
Number analyzed (Participants) | 9
Number analyzed (Tumors) | 12
participants | 0

2. Secondary Outcome: Audiologic Response
Description: Defined as improvement in speech discrimination score (SDS), defined as an improvement in the score above the 95% critical difference threshold, compared to baseline audiogram at initiation of treatment. Audiologic worsening: decrease in SDS score below the 95% critical difference threshold, compared to baseline audiogram at initiation of treatment.
  Patients with vestibular schwannomas will receive baseline audiograms within 28 days before enrollments and subsequent audiograms at the time of each MRI.
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 9
participants | 0

3. Primary Outcome: Change in Tumor Size From Baseline
Time Frame: 1 Year
Measure: Median (Full Range); unit: % of change in tumor size from baseline
Units Other Than Participants: Tumors
Arm/Group | RAD001
Number analyzed (Participants) | 9
Number analyzed (Tumors) | 12
% of change in tumor size from baseline | 5.72 [-14 to 25.71]

ADVERSE EVENTS:
Time Frame: Continuously throughout 1 year of study
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=10)
alkaline phosphatase increased (Investigations) | 2
anemia (Blood and lymphatic system disorders) | 5
anxiety (Psychiatric disorders) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1
AST increased (Investigations) | 3
azoospermia (Reproductive system and breast disorders) | 1
bruising (Injury, poisoning and procedural complications) | 1
chills (General disorders) | 1
cholesterol high (Investigations) | 7
constipation (Gastrointestinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
depression (Psychiatric disorders) | 1
diarrhea (Gastrointestinal disorders) | 4
dry skin (Skin and subcutaneous tissue disorders) | 3
dysgeusia (Nervous system disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
fatigue (General disorders) | 6
fever (General disorders) | 1
headache (Nervous system disorders) | 6
hyperglycemia (Metabolism and nutrition disorders) | 5
hypernatremia (Metabolism and nutrition disorders) | 5
hypertension (Vascular disorders) | 2
hypertriglyceridemia (Metabolism and nutrition disorders) | 4
hypoglycemia (Metabolism and nutrition disorders) | 1
hyponatremia (Metabolism and nutrition disorders) | 1
hypophosphatemia (Metabolism and nutrition disorders) | 2
irregular menstruation (Reproductive system and breast disorders) | 1
lymphocyte count decreased (Investigations) | 5
mucositis oral (Gastrointestinal disorders) | 10
muscle weakness- right sided (Musculoskeletal and connective tissue disorders) | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
neck pain (Musculoskeletal and connective tissue disorders) | 1
neutrophil count decreased (Investigations) | 3
non-cardiac chest pain (General disorders) | 1
pain (to bone; right clavicula) (Musculoskeletal and connective tissue disorders) | 1
pain (to extremity; left 4th finger) (Musculoskeletal and connective tissue disorders) | 1
pain (to right flank) (Musculoskeletal and connective tissue disorders) | 1
platelet count decreased (Investigations) | 6
pruritis (Skin and subcutaneous tissue disorders) | 4
rash (Skin and subcutaneous tissue disorders) | 5
rash acneiform (Skin and subcutaneous tissue disorders) | 1
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
scalp pain (Skin and subcutaneous tissue disorders) | 1
skin infection (Infections and infestations) | 1
toothache (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 1
white blood cell decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes